CLINICAL TRIAL: NCT05078866
Title: A Phase Ib/II Clinical Trial of Nous-209 for Recurrent Neoantigen Immunogenicity and Cancer Immune Interception in Lynch Syndrome
Brief Title: Cancer Preventive Vaccine Nous-209 for Lynch Syndrome Patients
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2021-10799; NCI-2021-10799 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2022-0065 (Other: M D Anderson Cancer Center); MDA21-06-01 (Other: DCP); P30CA016672 (NIH); UG1CA242609 (NIH)
Record Dates: First submitted 2021-10-14; First posted 2021-10-15 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Carcinoma; Lynch Syndrome
MeSH Terms: conditions — Colorectal Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Specimen Handling; Endoscopic Mucosal Resection; Endoscopy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part I (GAd20-209-FSPs, MVA-209-FSPs) (Experimental): Patients receive GAd20-209-FSPs IM on day 1 and MVA-209-FSPs IM at week 8. Patients undergo endoscopy with biopsy during screening and follow up as well as blood sample collection on the trial.
  Interventions: Biological: Adenoviral Tumor-specific Neoantigen Priming Vaccine GAd-209-FSP; Procedure: Biospecimen Collection; Procedure: Endoscopic Biopsy; Biological: MVA Tumor-specific Neoantigen Boosting Vaccine MVA-209-FSP; Other: Questionnaire Administration
- Part II Arm A (GAd20-209-FSPs, MVA-209-FSPs) (Experimental): Patients receive GAd20-209-FSPs IM at week 52 and MVA-209-FSPs IM at week 60. Patients undergo endoscopy with biopsy as well as blood sample collection on the trial.
  Interventions: Biological: Adenoviral Tumor-specific Neoantigen Priming Vaccine GAd-209-FSP; Procedure: Biospecimen Collection; Procedure: Endoscopic Biopsy; Biological: MVA Tumor-specific Neoantigen Boosting Vaccine MVA-209-FSP; Other: Questionnaire Administration
- Part II Arm B (MVA-209-FSPs) (Experimental): Patients receive MVA-209-FSPs IM at week 52. Patients undergo endoscopy with biopsy as well as blood sample collection on the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Endoscopic Biopsy; Biological: MVA Tumor-specific Neoantigen Boosting Vaccine MVA-209-FSP; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Adenoviral Tumor-specific Neoantigen Priming Vaccine GAd-209-FSP — Given IM
  Other Names: GAd-209-FSP; GAd20-209-FSP; Great Ape Adenoviral Tumor-specific Neoantigen Priming Vaccine GAd-209-FSP
  Arms: Part I (GAd20-209-FSPs, MVA-209-FSPs); Part II Arm A (GAd20-209-FSPs, MVA-209-FSPs)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Endoscopic Biopsy — Undergo endoscopy with biopsy
  Other Names: Endoscopy and Biopsy
Biological: MVA Tumor-specific Neoantigen Boosting Vaccine MVA-209-FSP — Given IM
  Other Names: Modified Vaccinia Ankara Tumor-specific Neoantigen Boosting Vaccine MVA-209-FSP; Modified Vaccinia Virus Ankara Tumor-specific Neoantigen Boosting Vaccine MVA-209-FSP; MVA-209-FSP
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase Ib/II trial evaluates the safety and effect of the Nous-209 vaccine in Lynch syndrome patients. Lynch syndrome is an inherited disorder in which affected individuals have a higher-than-normal chance of developing colorectal cancer and certain other types of cancer, often before the age of 50. In Lynch syndrome, errors in the genetic information inside cells are not properly corrected. When that happens, the cells produce new proteins called neoantigens. Neoantigens are recognized by the body's immune system as foreign, and the body tries to get rid of them. Nous-209 is a vaccine made with man-made copies of some of those neoantigens. This trial aims to see whether the Nous-209 vaccine is safe to give to patients with Lynch syndrome, whether people are able to take the Nous-209 vaccine without becoming too uncomfortable, and how the immune system of patients with Lynch syndrome respond to the Nous-209 vaccine. This trial may help researchers determine whether receiving Nous-209 have an effect on the development of polyps or tumors in the colon.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of adenoviral tumor-specific neoantigen priming vaccine GAd-209-FSP (GAd20-209-FSPs) (1 prime) and MVA tumor-specific neoantigen boosting vaccine MVA-209-FSP (MVA-209-FSPs) (1 boost) vaccination when administered as a single agent (monotherapy) in participants with Lynch syndrome (LS).

II. To evaluate the neoantigen-specific immunogenicity of GAd20-209-FSPs (1 prime) and MVA-209-FSPs (1 boost) vaccination when administered as a single agent (monotherapy) in participants with LS.

III. To evaluate the neoantigen-specific immunogenicity of GAd20-209-FSP prime and MVA-209-FSP boost or MVA-209-FSP boost alone when administered to previously-vaccinated immunogenic participants with LS.

IV. To evaluate the safety and tolerability of GAd20-209-FSP prime and MVA-209-FSP boost or MVA-209-FSP boost alone when administered to previously vaccinated immunogenic participants with LS.

SECONDARY OBJECTIVES:

I. To assess the effect of Nous-209 vaccination on T cell immune profile and T cell receptor (TCR) repertoire in the peripheral blood of participants with LS.

II. To assess the effect of Nous-209 vaccination on TCR repertoire within histologically normal colorectal mucosal of participants with LS.

III. To evaluate the effect of Nous-209 vaccination on tumor infiltrating lymphocyte (TIL) immune profile and TCR repertoire within colorectal adenomas in participants with LS.

IV. To assess the cytotoxicity of matched T cells on participant-derived colorectal adenoma organoids following Nous-209 vaccination in participants with LS.

V. To evaluate the effect of Nous-209 vaccination on the burden of colorectal adenomas/advanced neoplasia/carcinoma in participants with LS.

VI. To assess the effect of Nous-209 vaccination on the burden of LS-related carcinomas in participants with LS.

VII. To evaluate the effect of Nous-209 vaccination on cell free deoxyribonucleic acid (DNA) (cfDNA) mutation profiles and cfDNA burden in participants with LS.

VIII. To correlate tobacco and alcohol consumption with the immune response to Nous-209 in trial participants.

IX. To assess the mismatch repair (MMR) and/or microsatellite instability (MSI) status of polyps (and adjacent normal mucosa as control) detected in the baseline and end-of-the-study colonoscopy using different technologies such as immunohistochemistry, MSI analysis by polymerase chain reaction (PCR), or next-generation sequencing.

OUTLINE:

PART I: Patients receive GAd20-209-FSPs intramuscularly (IM) on day 1 and MVA-209-FSPs IM at week 8. Patients undergo endoscopy with biopsy during screening and follow up as well as blood sample collection on the trial.

PART II: Eligible patients from Part I are randomized to 1 of 2 arms.

ARM A: Patients receive GAd20-209-FSPs IM at week 52 and MVA-209-FSPs IM at week 60. Patients undergo endoscopy with biopsy as well as blood sample collection on the trial.

ARM B: Patients receive MVA-209-FSPs IM at week 52. Patients undergo endoscopy with biopsy as well as blood sample collection on the trial.

After completion of study treatment, patients are followed up at weeks 16, 24, 36, and 52.

ELIGIBILITY:
Inclusion Criteria:

* INCLUSION CRITERIA FOR PARTICIPANTS IN COHORT 1:
* Participants must have a clinical diagnosis of Lynch syndrome (LS) as defined by:

  * Mutation-positive LS: documented carriers (or obligate carriers by pedigree) of a germline mutation in MMR genes (MLH1, MSH2/EPCAM, MSH6, or PMS2) that is deleterious/pathogenic or suspected to be deleterious/pathogenic (known or predicted to be detrimental/loss of function, respectively). The mutation must have been identified through a Clinical Laboratory Improvement Act (CLIA)-approved laboratory setting or an equivalent international agency. Final determination of eligibility for any discordant results in pathogenicity of the mutation will be determined by the study investigator. A formal eligibility exception in those instances will not be required as long as approval by the overall study principal investigator (PI) has been granted and documented
  * Mutation-negative LS (also known as "Lynch-like syndrome" or "suspected Lynch syndrome): individuals with both of the following:

    * A personal history of a non-sporadic MMR-deficient premalignant lesion (i.e., colorectal polyp) or a non-sporadic MMR-deficient malignant tumor, where "non-sporadic MMR deficiency" is defined by (1) the loss of MLH1, MSH2, MSH6, or PMS2 expression by immunohistochemistry (IHC), or (2) the detection of MSI by PCR or both, but no evidence of MLH1 promoter methylation in cases with loss of both MLH1 and PMS2, All testing must have been performed in accordance with local institutional guidelines in a CLIA- approved setting. (Note: central confirmation of MMR expression status, MSI, MLH1 promoter methylation or BRAF mutation is not required.); and
    * Documented results of germline mutation testing performed in a CLIA-approved laboratory environment, demonstrating either a variant of unknown significance in MMR genes or the lack of a clinically significant variant in MMR genes; or, documentation that the individual declined to undergo germline MMR genetic testing
* Participants must have no evidence of active or recurrent invasive cancer for 6 months prior to screening
* Participants must be at least 6 months from any prior cancer-directed treatment (such as surgical resection, chemotherapy, immunotherapy, hormonal therapy, or radiation)
* Participants must have endoscopically accessible distal colon and/or rectal mucosa (i.e., participants must have at least part of the descending/sigmoid colon and/or rectum intact)
* Participants must consent to standard of care surveillance with colonoscopy with biopsies every 12 months
* Participants must consent to refrain from using aspirin or non-steroidal anti-inflammatory drugs (NSAIDs) or cyclooxygenase (COX) inhibitors for the duration of the trial, except for cardio-preventive aspirin (< 100 mg daily). Individuals taking such drugs may not be enrolled unless they are willing to stop the medications (and possibly change to alternative non-excluded medications to treat the same conditions) no less than 1 month prior to enrollment. Participants will discuss with their primary care provider/local provider about the discontinuation of such medication(s) and obtain approval prior to stopping any agent
* Age >= 18 years. Because no dosing or adverse event (AE) data are currently available on the use of Nous-209 in participants < 18 years of age, children are excluded from this study but will be eligible for future pediatric trials, if applicable
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Hemoglobin >= 10 g/dL or hematocrit >= 30 %
* Leukocyte count >= 3,500/microliter
* Platelet count >= 100,000/microliter
* Absolute neutrophil count >= 1,500/microliter
* Estimated glomerular filtration rate (eGFR) (or creatinine clearance calculated using the Cockcroft-Gault equation) ≥ 60 mL/min/1.73m^2 (mL/min, within institutional limits of normal)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2 times the institutional upper limit of normal (ULN)
* Total bilirubin =< 1.5 the ULN; participants with Gilbert's disease may be enrolled with higher total bilirubin if their direct bilirubin is =< 1.5 times the ULN
* Participants must consent to refrain from receiving any other type of vaccination during the first 10 weeks of the trial
* Participants must consent to refrain from receiving adenoviral-based vaccines for the duration of the trial (including the period from week 9 to week 52)
* Willing and able to adhere to the prohibitions and restrictions specified in the final approved protocol
* The effects of Nous-209 on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry for the duration of study participation (12 months) and 6 months after end of study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Ability to understand and the willingness to sign a written informed consent document (available for both English- and Spanish-speaking individuals)
* INCLUSION CRITERIA FOR PARTICIPANTS IN COHORT 2:
* Participants must have been confirmed eligible and met all study inclusion criteria for participation in study Cohort 1
* Participants must have completed all baseline procedures and received a complete cycle of GAd20- 209 FSP (prime) and MVA-209-FSP (boost) vaccination per protocol for Cohort 1
* Participants must have undergone collection of research blood samples at baseline (week 0) and week 9 for evaluation of the Nous-209-induced immunogenicity endpoint as specified for Cohort 1. Only participants with evaluable and proved immunogenicity response at Week 9 are eligible for participation in Cohort 2
* Participants must consent to refrain from receiving any other type of vaccination during weeks 52 to 68 of the trial
* Participants must consent to refrain from receiving adenoviral-based vaccines for the duration of the trial (including the period from week 52 to week 68)
* Participants must consent to refrain from using aspirin or non-steroidal anti-inflammatory drugs (NSAIDs) or cyclooxygenase (COX) inhibitors for the duration of the cohort 2, except for cardiopreventive aspirin (< 100 mg daily). Individuals taking such drugs may not be enrolled unless they are willing to stop the medications (and possibly change to alternative non-excluded medications to treat the same conditions) no less than 1 month prior to enrollment. Participants will discuss with their primary care provider/local provider about the discontinuation of such medication(s) and obtain approval prior to stopping any agent
* Female participant must agree to a pregnancy test at week 52

Exclusion Criteria:

* Prior receipt of a recombinant adenoviral or MVA vaccine including COVID-19 adenovirus vaccines within the previous 6 months
* Histologically-confirmed high-grade dysplasia or cancer on biopsy at screening
* Individuals with active malignancy (excluding non-melanoma skin cancer)
* Any serious uncontrolled and/or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with participant's safety, obtaining informed consent, or compliance to the study procedures
* Active infection (acute and self-limited) or human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection. Participants with laboratory evidence of cleared HBV and HCV infection will be permitted
* History of organ allograft or other history of immunodeficiency
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to study drug, or excipients, or to egg proteins
* Individuals with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications (such as infliximab, rituximab, adalimumab, tacrolimus) within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Pregnant or breastfeeding or planning to become pregnant within 6 months after the end of study. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with Nous-209, breastfeeding should be discontinued if the mother is treated with Nous-209
* Men attempting or planning to conceive children during the study or within 6 months after the end of the study
* Participants may not be receiving any other investigational agents
* Cohort 2 only: participants who experienced grade 3 or higher AEs attributed to study drug in Cohort 1, excluding reactogenicity events

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Rates of grade 2/3 adverse events and symptom reactivity following vaccination | Up to 12 months
Rate of immunogenicity following vaccination (Cohort I) | Baseline and week 9
  Immunogenicity will be defined as reactivity to at least 1 of 16 synthetic FSP pools using an enzyme-linked immune absorbent spot (ELISpot) assay. The rate of immunogenicity induced by Nous-209 will be reported along with its 95% exact (Clopper-Pearson) confidence interval.
Rate of immunogenicity following revaccination (Cohort II) | Weeks 52 and at 8 weeks after the last boost with MVA-209-FSP (corresponding to week 68 and week 60, for arm A and B, respectively)
  Immunogenicity will be defined as reactivity to at least 1 of 16 synthetic FSP pools using an enzyme-linked immune absorbent spot (ELISpot) assay. The rate of immunogenicity induced by Nous-209 will be reported along with its 95% exact (Clopper-Pearson) confidence interval.
Rates of grade 2/3 adverse events and symptom reactivity following revaccination (Cohort II) | Up to 12 months

SECONDARY OUTCOMES:
Changes in T cell immune profile and T cell receptor (TCR) repertoire in the peripheral blood | Baseline up to 12 months
Changes in TCR repertoire within histologically normal colorectal mucosal | Baseline to 12 months
Changes in the gene expression profile and TCR repertoire of tumor infiltrating lymphocytes (TIL) within colorectal adenomas | Baseline to 12 months
T cell cytotoxicity against matched colorectal adenoma organoids | At 12 months
Percentage change in the number of colorectal adenomas, advanced neoplasia, and/or carcinomas | At 12 months
  Will use two-sample t-test and general linear models for the comparison.
Rate of Lynch syndrome-related carcinomas | At 12 months
Change in cell free deoxyribonucleic acid (cfDNA) detectability and mutation profile in the peripheral blood | Baseline up to 12 months
Immune response to Nous-209 | Up to 12 months
  Tobacco and alcohol consumption will be correlated with the immune response to Nous-209 in trial participants.
Mismatch repair and/or microsatellite instability status of polyps (and adjacent normal mucosa as control) | Baseline to 12 months
  Will be assessed using different technologies such as immunohistochemistry, MSI analysis by polymerase chain reaction, or next-generation sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Vilar-Sanchez, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (3):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
- University of Puerto Rico, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] D'Alise AM, Willis J, Duzagac F, Hall MJ, Cruz-Correa M, Idos GE, Thirumurthi S, Ballester V, Leoni G, Garzia I, Antonucci L, De Marco L, Micarelli E, Deng N, Secli L, Gogov S, Dong W, Jack Lee J, Bowen CM, Vornik LA, Garcia-Gonzalez A, Reyes-Uribe L, Richmond E, Umar A, Brown PH, Sinha KM, Rodriguez LM, Scarselli E, Vilar E. Nous-209 neoantigen vaccine for cancer prevention in Lynch syndrome carriers: a phase 1b/2 trial. Nat Med. 2026 Jan 16. doi: 10.1038/s41591-025-04182-9. Online ahead of print. PMID 41545594

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT05078866/Prot_SAP_000.pdf